CLINICAL TRIAL: NCT05639023
Title: The Orthopaedic Manipulation Techniques of the Lin School of Lingnan Region in the Treatment of Adolescent Idiopathic Scoliosis - A Randomized Controlled Study
Brief Title: Orthopaedic Manipulation in Treatment of Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kiu Lam Chung, Associate Professor of Practice in Chinese Medicine, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.353
Record Dates: First submitted 2022-10-26; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manipulation Techniques Group (Experimental): Subjects will be received orthopedic manipulation and Physiotherapy Scoliosis-Specific Exercise(PSSE). For orthopedic manipulation, Subjects will received 12 times orthopedic manipulation. Three times of treatment per months, and less than twice a week. For PSSE, subjects will receive 14 supervise training, 5 times of intensive supervise training for first two weeks and then 1-2 trainings per month for the rest. Subjects are encouraged to perform home exercise everyday on their own throughout the study.
  Interventions: Other: Manipulation Techniques; Other: Physiotherapy Scoliosis-Specific Exercise
- Control Group (Experimental): Subjects will be received sham orthopedic manipulation and Physiotherapy Scoliosis-Specific Exercise(PSSE). For orthopedic manipulation, Subjects will received 12 times orthopedic manipulation. Three times of treatment per months, and less than twice a week. For PSSE, subjects will receive 14 supervise training, 5 times of intensive supervise training for first two weeks and then 1-2 trainings per month for the rest. Subjects are encouraged to perform home exercise everyday on their own throughout the study.
  Interventions: Other: Physiotherapy Scoliosis-Specific Exercise

INTERVENTIONS:
Other: Manipulation Techniques — Subjects will received 12 times orthopedic manipulation. Three times of treatment per months, and less than twice a week.
  Arms: Manipulation Techniques Group
Other: Physiotherapy Scoliosis-Specific Exercise — Subjects will receive 14 supervise training, 5 times of intensive supervise training for first two weeks and then 1-2 trainings per month for the rest. Subjects are encouraged to perform home exercise everyday on their own throughout the study.

SUMMARY:
To examine the clinical efficacy of the Orthopaedic Manipulation Techniques of the Lin School of Lingnan Region in the treatment of Adolescent Idiopathic Scoliosis

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent will undergo a 0-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a single-blind manner(participant) in a 1:1 ratio to Manipulation Techniques Group or Control Group.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged between 10 and 18 who can speak and read Chinese
2. Fulfil the diagnostic criteria of scoliosis, i.e. Cobb's angle ≥ 10 degree
3. Risser grade ranging from 0 to 4
4. Informed consent agreement signed by both subject and their parents/guardians
5. Able to participate in follow-up assessments

Exclusion Criteria:

1. History of spine surgery;
2. Cobb's angle >30 degrees
3. Known to have severe respiratory or cardiovascular comorbidities; vertebral tumours and spinal canal abnormalities; Leukaemia, thrombocytopenia and other bleeding disorders
4. Known to have cognitive impairment.
5. Documented pregnancy
6. Wearing brace within 1 month.
7. Involved in other interventional clinical studies at the same time.
8. Uncooperative during treatments
9. Being assessed by investigators as unsuitable to participate.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-19 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of Scoliosis Research Society-22 (SRS-22) | Baseline, Week 8,16,24
  Scoliosis Research Society-22 (SRS-22) questionnaire includes 5 dimensions : 1)function/activity,2) pain,3) self-perceived image, 4)mental health, satisfaction with treatment and 5)other health-related quality of life(HRQL) parameters with a total of 22 items, and is scored by the Likert 5-level scoring method. Possible score range from 0 (no pain)to 5(worst possible pain).A higher score indicates a better quality of life for the patient.

SECONDARY OUTCOMES:
Change of Traditional Chinese version of Spinal Appearance Questionnaire score (TC-SAQ) | Baseline, Week 8,16,24
  Spinal Appearance Questionnaire (SAQ) is a questionnaire specifically assess the cosmetic perception of AIS patients. The reliability, validity and responsiveness of SAQ have been demonstrated to be excellent for the assessment of appearance in AIS patients
Change of Cobb's angle measured by Xray | Baseline, Week 16
  A standing whole-spine PA radiograph will be used for measurement. The measurement method is: 1) identify the most inclined vertebrae in the superior section and draw a perpendicular line. Then, 2) identify the most inclined vertebrae in the inferior section and 3) draw a perpendicular line. The angle formed at the intersection of these two lines is the Cobb's angle.
Change of spinal rotation by Ultrasonography | Before and after the manipulation with the duration of 16 weeks
  Scolioscan is a validated radiation-free system for scoliosis assessment in clinics by using coronal images of spine generated by a 3D ultrasound volume projection imaging method. Scolioscan Air, a portable device of developed from Scolioscan, can be used to monitor the spinal development during study
Change of muscle volume by Ultrasonography | Before and after every manipulation with the treatment duration of 16 weeks
  Scolioscan is a validated radiation-free system for scoliosis assessment in clinics by using coronal images of spine generated by a 3D ultrasound volume projection imaging method. Scolioscan Air, a portable device of developed from Scolioscan, can be used to monitor the spinal development during study
Change of Cobb's angle measured by Ultrasonography | Before and after the manipulation with the duration of 16 weeks
  Scolioscan is a validated radiation-free system for scoliosis assessment in clinics by using coronal images of spine generated by a 3D ultrasound volume projection imaging method. Scolioscan Air, a portable device of developed from Scolioscan, can be used to monitor the spinal development during study

REFERENCES:
- [Derived] Hung HY, Kong WC, Tam TH, Leung PC, Zheng Y, Wong AYL, Lin Z, Yao F, Tian Q, Mok TL, Loo LE, Chung KL. Efficacy and safety of the orthopaedic manipulation techniques of the Lin School of Lingnan Region in the treatment of adolescent idiopathic scoliosis: protocol of a participant-and-assessor-blinded randomized controlled study. BMC Musculoskelet Disord. 2024 Jan 4;25(1):32. doi: 10.1186/s12891-023-07152-9. PMID 38178051